CLINICAL TRIAL: NCT03928522
Title: Prospective Randomized Study Investigating the Characterization of Antibiotics From Antibiotic Impregnated Cement After Total Knee Arthroplasty
Brief Title: Antibiotic Elution in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201811101
Record Dates: First submitted 2019-01-29; First posted 2019-04-26 (Actual); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Total Knee Replacement
MeSH Terms: interventions — Vancomycin; Tobramycin

STUDY DESIGN:
Who Masked: Participant
Masking Description: patient will not know which antibiotic cement group they are in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Pre-mixed tobramycin (Active Comparator): patients will receive pre-mixed tobramycin cement
  Interventions: Device: pre-mixed tobramycin
- hand mixed tobramycin (Active Comparator): patients will receive hand mixed tobramycin cement
  Interventions: Drug: hand mixed tobramycin
- hand mixed vancomycin (Active Comparator): patients will receive hand mixed vancomycin cement
  Interventions: Drug: hand mixed vancomycin
- hand-mixed vancomycin and tobramycin (Experimental): patients will receive hand mixed vancomycin and tobramycin
  Interventions: Drug: hand mixed vancomycin; Drug: hand mixed tobramycin

INTERVENTIONS:
Drug: hand mixed vancomycin — hand mixed vancomycin powder into cement
  Other Names: Vancomycin
  Arms: hand mixed vancomycin; hand-mixed vancomycin and tobramycin
Drug: hand mixed tobramycin — hand mixed tobramycin into cement
  Other Names: Tobramycin
  Arms: hand mixed tobramycin; hand-mixed vancomycin and tobramycin
Device: pre-mixed tobramycin — this cement is already pre-mixed with tobramycin
  Other Names: Antibiotic PMMA bone cement
  Arms: Pre-mixed tobramycin

SUMMARY:
The purpose of the study is to characterize and quantify the level of antibiotics eluted from antibiotic laden cement after primary cemented total knee arthroplasty.

Patients will be identified by medical record review to make sure they meet inclusion and exclusion criteria.

Patients that qualify and sign consent will be randomized to 1 of 4 antibiotic cement groups which are pre-mixed tobramycin, hand-mixed tobramycin, hand mixed vancomycin, and hand-mixed tobramycin and hand mixed vancomycin. Study patients will be blinded to their study group. Intraoperative fluid from the knee prior to surgery and postoperative drain fluid from the knee postoperatively will be collected as well.

DETAILED DESCRIPTION:
Patients will be identified by medical record review to make sure they meet inclusion and exclusion criteria.

Patients that qualify and sign consent will be randomized to 1 of 4 antibiotic cement groups which are pre-mixed tobramycin, hand-mixed tobramycin, hand mixed vancomycin, and hand-mixed tobramycin and hand mixed vancomycin. Study patients will be blinded to their study group. Intraoperative fluid from the knee prior to surgery and postoperative drain fluid from the knee postoperatively will be collected as well.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Total knee arthroplasty for primary osteoarthritis performed by Dr. Rick Wright.
* Primary diagnosis of knee osteoarthritis

  * Exclusion Criteria:
* Diminished mental capacity
* Vancomycin allergy
* Tobramycin allergy
* Patient history requiring IV administration of vancomycin or tobramycin perioperatively
* Chronic kidney disease stage III and stage IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Lawrie, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Orthopedics, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intra-articular Vancomycin: Patients will receive powdered vancomycin antibiotic into a cementless total knee in wound prior to closure
Period: Overall Study
Arm/Group | Pre-mixed Tobramycin | Hand Mixed Tobramycin | Hand Mixed Vancomycin | Hand-mixed Vancomycin and Tobramycin | Intra-articular Vancomycin
Started | 12 | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intr-articular Vancomycin: Patients will receive powdered vancomycin antibiotic into a cementless total knee in wound prior to closure
- Total: Total of all reporting groups
Arm/Group | Pre-mixed Tobramycin | Hand Mixed Tobramycin | Hand Mixed Vancomycin | Hand-mixed Vancomycin and Tobramycin | Intr-articular Vancomycin | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 6 | 3 | 7 | 23
  >=65 years | 8 | 9 | 6 | 9 | 5 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 6 | 6 | 7 | 31
  Male | 4 | 8 | 6 | 6 | 5 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 12 | 12 | 60

OUTCOME MEASURES:

1. Primary Outcome: Amount of Vancomycin and Tobramycin Eluted From Hand Mixed Cement With Both Antibiotics After Total Knee Arthroplasty
Description: We wanted to measure the effect of elution level of vancomycin and tobramycin together
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: mg/mL
Arm/Group | Pre-mixed Tobramycin | Hand Mixed Tobramycin | Hand Mixed Vancomycin | Hand-mixed Vancomycin and Tobramycin | Intr-articular Vancomycin
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
mg/mL | 23.9 [9.8 to 125.4] | 30.6 [8.6 to 81.0] | 12.6 [2.0 to 72.6] | 16.2 [.3 to 47.3] | 1315 [429 to 2324.8]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected within 4-6 weeks after surgery.
Groups:
- Intra-articular Vancomycin: patients will receive powdered vancomycin into the wound before closure
Arm/Group | Pre-mixed Tobramycin | Hand Mixed Tobramycin | Hand Mixed Vancomycin | Hand-mixed Vancomycin and Tobramycin | Intra-articular Vancomycin
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT03928522/Prot_SAP_001.pdf